CLINICAL TRIAL: NCT04028050
Title: A Phase IIIB, Single Arm, Multicenter Study of Atezolizumab (Tecentriq) in Combination With Carboplatin Plus Etoposide to Investigate Safety and Efficacy in Patients With Untreated Extensive-Stage Small Cell Lung Cancer - MAURIS
Brief Title: A Study of Atezolizumab in Combination With Carboplatin Plus Etoposide to Investigate Safety and Efficacy in Patients With Untreated Extensive-Stage Small Cell Lung Cancer
Acronym: MAURIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML41118
Record Dates: First submitted 2019-07-19; First posted 2019-07-22 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Small Cell Lung Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — atezolizumab; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atezolizumab + Carboplatin + Etoposide (Experimental): Participants will receive intravenous infusions of atezolizumab 1200 milligrams (mg) in combination with carboplatin to achieve an initial target area under the concentration-time curve (AUC) of 5 milligrams per milliliter per minute (mg/mL/min), followed by intravenous infusion of etoposide 100 milligrams per square meter (mg/m^2) on days 1 through 3 of each cycle during the induction phase (21-day cycle for four/six cycles). On Days 2 and 3, participants will receive etoposide alone. After the induction phase, participants will begin maintenance therapy with atezolizumab every 3 weeks until PD, unacceptable toxicity, loss of clinical benefit or study termination by the Sponsor.
  Interventions: Drug: Atezolizumab; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered by IV infusion at a fixed dose of 1200 mg on Day 1 of each 21-day cycle until unacceptable toxicity or loss of clinical benefit as determined by the investigator. After the induction phase, participants will begin maintenance therapy with atezolizumab every 3 weeks.
  Other Names: MPDL3280A, RO5541267, Tecentriq
Drug: Carboplatin — Carboplatin will be administered after completion of atezolizumab by IV infusion over 30-60 minutes to achieve an initial target AUC of 5 mg/mL/min (Calvert formula dosing) with standard anti-emetics per local practice guidelines.
Drug: Etoposide — Etoposide will be administered by IV infusion over 60 minutes following carboplatin administration, during the induction phase on Day 1 through 3 of each cycle. On Days 2 and 3, patients will receive etoposide alone.

SUMMARY:
This is a phase IIIB, single-arm, single-country, multicenter study of the safety and efficacy of atezolizumab in combination with carboplatin plus etoposide in patients who have ES-SCLC and are chemotherapy-naive for their extensive-stage disease.

DETAILED DESCRIPTION:
Induction treatment will be administered on a 21-day cycle for four/six cycles. Following the induction phase, participants will continue maintenance therapy with atezolizumab. Maintenance with atezolizumab will continue until disease progression (PD), unacceptable toxicity or loss of clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed ES-SCLC per the Veterans Administration Lung Study Group (VALG) staging system
* Measurable disease, as defined by RECIST v1.1. Previously irradiated lesions can only be considered as measurable disease if disease progression has been unequivocally documented at that site since radiation and the previously irradiated lesion is not the only site of disease
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) from 0 to 2
* Life expectancy > 12 weeks
* No prior systemic treatment for ES-SCLC
* Patients who have received prior chemoradiotherapy for limited-stage SCLC must have been treated with curative intent and experienced a treatment-free interval of at least 6 months since last chemotherapy, radiotherapy, or chemoradiotherapy cycle from diagnosis of ES-SCLC
* Patients where thoracic radiotherapy (consolidation RT) is clinically indicated could be enrolled providing they receive RT between the completion of induction phase and the beginning of maintenance phase
* Patients with Paraneoplastic syndromes can be enrolled if an autoimmune origin can be excluded
* Adequate hematologic and end organ function
* Negative human immunodeficiency virus (HIV) test at screening
* Negative hepatitis B surface antigen (HBsAg) test at screening
* Negative total hepatitis B core antibody (HBcAb) test at screening, or positive total HBcAb test followed by a negative hepatitis B virus (HBV) DNA test at screening
* Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening. The HCV RNA test will be performed only for patients who have a positive HCV antibody test.
* For women of childbearing potential: agreement to remain abstinent or use of contraception
* For men: agreement to remain abstinent or use a condom, and agreement to refrain from donating sperm

Exclusion Criteria:

* Symptomatic or actively progressing central nervous system (CNS) metastases. Asymptomatic patients with treated or untreated CNS lesions are eligible, provided that all of the following criteria are met: (1) Measurable disease, per RECIST v1.1, must be present outside the CNS. (2) Patient has no history of intracranial hemorrhage or spinal cord hemorrhage. (3) Patient has not undergone stereotactic radiotherapy within 7 days prior to initiation of study treatment, whole-brain radiotherapy within 14 days prior to initiation of study treatment, or neurosurgical resection within 28 days prior to initiation of study treatment. (4) Patient has no ongoing requirement for corticosteroids as therapy for CNS disease. Anticonvulsant therapy at a stable dose is permitted. Metastases are limited to the cerebellum or the supratentorial region. (5) There is no evidence of interim progression between completion of CNS directed therapy and initiation of study treatment. (6) Asymptomatic patients with CNS metastases newly detected at screening are allowed at Investigator's discretion with no need to repeat the screening brain scan.
* History of leptomeningeal disease
* Uncontrolled tumor-related pain
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures. Patients with indwelling catheters are allowed regardless of drainage frequency.
* Uncontrolled or symptomatic hypercalcemia
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computerized tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Active tuberculosis
* Significant cardiovascular disease within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
* Major surgical procedure other than for diagnosis within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
* History of malignancy other than SCLC within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death, such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer
* Prior allogeneic stem cell or solid organ transplantation treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab
* Current treatment with anti-viral therapy for HBV
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within 5 months after the final dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2023-07-13 (Actual); Study Completion 2023-07-13 (Actual)

PRIMARY OUTCOMES:
Incidence of Serious Adverse Events | 4 weeks after last dose of study treatment
Incidence of Serious and Non-Serious Immune Mediated Adverse Events | 4 weeks after last dose of study treatment

SECONDARY OUTCOMES:
Overall Survival (OS) Rate at 1 Year | 1 Year
  OS at 1 year, defined as the proportion of participants remaining alive at 1 year after initiation of study treatment.
Overall Survival (OS) Rate at 2 Years | 2 Years
  OS at 2 years, defined as the proportion of participants remaining alive at 2 years after initiation of study treatment.
Overall Survival (OS) Rate at 3 Years | 3 Years
  OS at 3 years, defined as the proportion of participants remaining alive at 3 years after initiation of study treatment.
Overall Survival (OS) Rate | Up to approximately 54 months
  OS, defined as the time from initiation of study treatment to death from any cause
Progression-Free Survival (PFS) | Up to approximately 54 months
  PFS, defined as the time from initiation of study treatment to the first occurrence of disease progression or death from any cause, whichever occurs first. PFS will be calculated based on disease status evaluated by the investigator according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1)
Objective response rate (ORR) | Up to approximately 54 months
  ORR, defined as the percentage of patients who attain complete response (CR) or partial response (PR) according to RECIST v1.
Duration of Response (DOR) | Up to approximately 54 months
  Duration of response (DOR), defined as the time from initial response to disease progression or death among patients who have experienced a CR or PR (unconfirmed) during the study. Duration of response will be calculated based on disease status evaluated by the investigator according to RECIST v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (25):
- Italy (25):
  - Presidio Ospedaliero Vito Fazzi; Unita Operativa Di Oncologia Medica, Lecce, Apulia
  - Ist. Ricovero e Cura a Carattere Scientifico-Centro Rif. Oncologico della Basilica, Rionero in Vulture (PZ), Basilicate
  - Azienda Ospedaliera di Rilievo Nazionale e di Alta Specialita San Giuseppe Moscati, Avellino, Campania
  - Az. Osp. Monaldi; 2 Pneumologia-Chemioterapia E Day Hospital-Pneumoncologia, Napoli, Campania
  - Azienda Osp Uni Seconda Università Degli Studi Di Napoli; Unità Operativa Oncologia Medica, Napoli, Campania
  - Istituto Nazionale per lo Studio e la Cura dei Tumori Fondazione G. Pascale, Napoli, Campania
  - Azienda Ospedaliero-Universitaria S.Orsola-Malpighi; Unità Operativa Oncologia Medica, Bologna, Emilia-Romagna
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola; Oncologia Medica, Meldola, Emilia-Romagna
  - Centro Di Riferimento Oncologico; Struttura Operativa Complessa Di Oncologia Medica B, Aviano, Friuli Venezia Giulia
  - Policlinico Universitario Campus Biomedico; Uoc Oncologia Medica, Rome, Lazio
  - Policlinico Universitario Agostino Gemelli, Rome, Lazio
  - Azienda Ospedaliera San Camillo Forlanini, Rome, Lazio
  - ASL 3 Genovese, Genoa, Liguria
  - ASST Spedali Civili di Brescia, Brescia, Lombardy
  - Ospedale San Raffaele S.r.l., Milan, Lombardy
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy
  - Irccs Istituto Europeo di Oncologia (IEO); Divisione di Oncologia, Milan, Lombardy
  - A.O.U. Maggiore della Carità, Novara, Piedmont
  - Azienda Unita Sanitaria Locale N1 Sassari; Unita Operativa Di Oncologia Medica, Sassari, Sardinia
  - Azienda Ospedaliera Vincenzo Cervello, Palermo, Sicily
  - Ospedale San Vincenzo Taormina :Divisione di Oncologia Medica, Taormina, Sicily
  - Ospedali Riuniti Di Ancona; Oncology, Ancona, The Marches
  - Azienda Ospedaliera Universitaria Pisana - Ospedale Cisanello; Dipartimento Cardio Toraco Vascolare, Pisa, Tuscany
  - ULSS2 Marca Trevigiana; UOC Oncologia Medica - Distretto di Treviso, Treviso, Veneto
  - Azienda Ospedaliera Universitaria Integrata Verona; UOC Oncologia, Verona, Veneto

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Bria E, Morgillo F, Garassino MC, Ciardiello F, Ardizzoni A, Stefani A, Verderame F, Morabito A, Chella A, Tonini G, Gilli M, Del Signore E, Berardi R, Mencoboni M, Bearz A, Delmonte A, Migliorino MR, Gridelli C, Pazzola A, Iero M, De Marinis F. Atezolizumab Plus Carboplatin and Etoposide in Patients with Untreated Extensive-Stage Small-Cell Lung Cancer: Interim Results of the MAURIS Phase IIIb Trial. Oncologist. 2024 May 3;29(5):e690-e698. doi: 10.1093/oncolo/oyad342. PMID 38377176